CLINICAL TRIAL: NCT04952792
Title: Pharmacokinetics, Pharmacodynamics and Safety of Apixaban on Hemodiafiltration
Brief Title: Study of Apixaban in Patients Receiving Hemodiafiltration
Acronym: HEMOCIONA
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hospital Universitari de Bellvitge (Other)
Collaborators: Spanish Society of Nephrology (Other); Baxter Healthcare Corporation (Industry)
Responsible Party: Principal Investigator, MIGUEL HUESO VAL, Principal Investigator, Hospital Universitari de Bellvitge
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2018-002991-41
Record Dates: First submitted 2021-06-09; First posted 2021-07-07 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-09

CONDITIONS: Atrial Fibrillation; Hemodialysis Complication
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Apixaban (Experimental): Apixaban treatment, oral, 2.5 mg/12h, 28 days
  Interventions: Drug: Apixaban 2.5 milligram Oral Tablet

INTERVENTIONS:
Drug: Apixaban 2.5 milligram Oral Tablet — Apixaban 2.5mg/12h, oral, 28 days

SUMMARY:
Atrial fibrillation (AF) is a prevalent and serious disease in hemodialysis (HD) patients. Untreated AF increases the risk of deaths related to cardiovascular events and multiplies the risk of strokes by 5. Anticoagulation with warfarin significantly reduces the incidence of ischemic strokes in the general population, has a long half-life, and a narrow therapeutic index that requires periodic monitoring. In addition, warfarin treatment is a frequent cause of hospital admission for iatrogenesis. In HD patients, the relationship between stroke prevention benefit and bleeding risk is an unmet medical need. It should be noted that in these patients the risk of bleeding is multiplied by 3 to 10 times compared to the general population. The new direct-acting oral anticoagulants (NACOs), thrombin inhibitors (dabigatran), and activated factor X inhibitors (rivaroxaban, apixaban, edoxaban), do not require regular monitoring, but their plasma concentrations are altered with the deterioration of the renal function. According to its technical data sheets, they do not recommend its use in clinical practice for HD patients. However, the apixaban data sheet includes the results of a pilot clinical trial in the African American population on HD, suggesting that it is a safe anticoagulant drug.

The objective of this clinical trial is to evaluate the pharmacokinetics, pharmacodynamics, and short-term safety (4 weeks) of apixaban in the Spanish population with non-valvular atrial fibrillation and on hemodialysis.

Long-term safety will be assessed in the extension study: prospective cohort study of patients included in the clinical trial. Therefore, this project is comprised of 2 clinical studies (one clinical trial and one extension study) whose objective is to evaluate the pharmacokinetics, pharmacodynamics, and short and long-term safety of apixaban in patients on hemodialysis and with non-valvular atrial fibrillation (FANV).

The results of this project (clinical trial and extension study) will provide evidence on whether apixaban may be the anticoagulant treatment of choice for this type of patient.

DETAILED DESCRIPTION:
7.1 CURRENT STATUS OF SCIENTIFIC-TECHNICAL KNOWLEDGE Despite technological advances, cardiovascular disease remains the most frequent cause of death in hemodialysis (HD) patients. The higher prevalence of diabetes, anemia, hyperparathyroidism and hypertension in the population with chronic kidney disease (CKD) favors the appearance of cardiac structural lesions. In addition, hypervolemia and hydroelectrolytic abnormalities increase the risk of arrhythmias. In fact, the annual incidence of atrial fibrillation (AF) in the hemodialysis population is 15 times higher than the general population of the same age and the risk of presenting a thromboembolic complication by a 5-fold increase.

Safely reducing the risk of thromboembolism in patients with AF and CKD is an unmet medical need. Prospective studies conducted in patients with AF have been systematically excluded in patients with a Glomerular Filtration Rate (GFR) <30 ml / min. Importantly, patients with CKD have alterations in hemostasis that predisposes patients to bleeding (reduction of alpha granules in platelets, reduction of endothelial adhesion molecules) and thrombosis (increased fibrinogen). This makes it impossible to extrapolate data from the population with normal kidney function.

Oral anticoagulant treatment with cumarinics such as warfarin, drugs that act as vitamin K antagonists (AVK), have been shown to be effective in reducing the risk of stroke and mortality. However, these drugs are not exempt from major complications since it is difficult to maintain a stable therapeutic index (INR). This frequently leads to the appearance of hemorrhages (the risk is 2 times higher than in HD patients without anticoagulant treatment) due to its reduced therapeutic margin and numerous interactions with drugs and foods, which makes it difficult to predict the pharmacokinetics of these drugs. The use of anticoagulants in patients with AF and in HD is a controversial topic. For example, the Kidney Disease: Improving Global Outcomes (KDIGO2012) guidelines do not recommend its use, while the American College of Cardiology (ACC) / American Heart Association (AHA) / Heart Rhythm Society 2014 guidelines does recommend its use. A recent meta-analysis, which included 7 studies, concluded that warfarin does not reduce the number of strokes and, in addition, was associated with a greater number of hemorrhages. In summary, there is not enough high-quality evidence to recommend warfarin for stroke prevention in patients on hemodialysis with AF. Furthermore, AVKs favor vascular calcifications and have been related to calciphylaxis lesions, CKD-associated pathologies.

7.2. New oral anticoagulants. Apixaban New oral anticoagulants (DOACs) are currently available, such as direct inhibitors of thrombin (dabigatran) and activated factor X (rivaroxaban, apixaban, edoxaban). These drugs have demonstrated their clinical efficacy in patients with GFR> 25 mL/min. DOACs offer the advantage that monitoring of their plasma levels is not necessary. Importantly, administration of dabigatran and rivaroxaban in hemodialysis patients has been associated with an increased risk of bleeding and death compared to warfarin. In contrast, apixaban, a priori, would be the oral anticoagulant of choice in hemodialysis patients.

Apixaban is a direct, selective and reversible coagulation Factor Xa (FXa) inhibitor that is approved to reduce the risk of stroke and systemic embolism in patients with AF of nonvalvular origin without increasing the risk of bleeding. Apixaban has a rapid absorption, a half-life of 12 h, it is metabolized by cytochrome P450 and 25% is eliminated via the kidneys (the rest is eliminated via the digestive tract).

Pharmacokinetic and pharmacodynamic studies of apixaban in patients with severe chronic kidney disease (CrCr= 15 mL/min) and in Hemodialysis observed an increase in exposure (area under the curve of plasma concentration vs. time was 44% and 36% respectively). This increased exposure is directly correlated with increased anti-Factor Xa activity. However, no changes were observed in terms of t1/2 (12 hours), maximum concentration (Cmax) or the presence of adverse effects. In a standard conventional hemodialysis session, the exposure to apixaban is decreased by 14%. A subsequent study observed the trend towards stability of apixaban levels after the administration of a reduced dose of apixaban 2.5mg/12h for a week in a sustained manner, therefore it has been suggested that it can be used in HD without the need for modify the dose. It should be borne in mind that all the studies that have analyzed the behavior of apixaban in HD have been carried out in the African American population of the United States, where the use of convective techniques (HDF) that allow greater elimination of medium and high molecular weight and that can modify the behavior of drugs with strong binding to plasma proteins. Apixaban could be affected by this phenomenon as it is a drug with strong protein binding (UPP 86%). In Catalonia, 65% of patients are on renal replacement therapy with HDF..

According to the technical data sheet (Section 5.2. Pharmacokinetic properties), in patients with renal insufficiency: "renal insufficiency had no manifest effect on the relationship between plasma concentration and anti-Factor Xa activity of apixaban", and in patients with end-stage renal disease: "theArea under the Curve (AUC) of apixaban was increased by 36% compared to that observed in subjects with normal renal function, when a single 5mg dose of apixaban was administered immediately after hemodialysis. Hemodialysis, started 2 hours after administration of a single 5mg dose of apixaban, decreased the AUC by 14% in these CKD subjects, corresponding to an apixaban clearance of 18 mL/min during hemodialysis. Therefore, hemodialysis is unlikely to be an effective measure to manage apixaban overdose." Apixaban appears to be a safe anticoagulant in hemodialysis patients. It should be noted that this study was conducted in the African American population (87.5%), so we do not know if these data could be extrapolated to the Spanish population. Apixaban was marketed in May 2011 and is indicated for "the prevention of stroke and systemic embolism in adult patients with nonvalvular atrial fibrillation (NVAF) with one or more risk factors such as stroke or previous transient ischemic attack (TIA); age ≥75 years; hypertension; mellitus diabetes; symptomatic heart failure (NYHA scale: ≥2). However, there is no information on the modification of its efficacy with the type of hemodialysis technique, and therefore if it could be used in clinical practice in hemodialysis patients.

7.3. Work Hypothesis

1. Apixaban is a safe oral anticoagulant in patients in our setting with chronic kidney disease (undergoing hemodiafiltration or hemodialysis) and nonvalvular atrial fibrillation.
2. Considering that severe renal dysfunction increases the AUC of apixaban by 36% and hemodialysis treatment only decreases exposure to the drug by 14%, the recommended dose of apixaban for patients on hemodialysis or hemodiafiltration is 2.5 mg/12h.
3. Apixaban is an effective oral anticoagulant in patients in our setting with chronic kidney disease (being treated with hemodiafiltration or hemodialysis) and nonvalvular atrial fibrillation:

   1. Plasma apixaban concentrations are stable in patients in our setting with chronic kidney disease (undergoing hemodiafiltration or hemodialysis) and nonvalvular atrial fibrillation.
   2. The anti-Factor Xa activity of apixaban is not affected in patients in our setting with chronic kidney disease (being treated with hemodiafiltration or hemodialysis) and nonvalvular atrial fibrillation.

ELIGIBILITY:
Inclusion Criteria:

Adults (18 years or older).

* Body weight ≥ 60 kg.
* Diagnosis of chronic kidney disease on hemodialysis, clinically stable (with a minimum of 3 months of treatment) and nonvalvular atrial fibrillation in treatment with coumarins.
* Patient candidate for change of anticoagulant treatment.
* In women of childbearing age, negative pregnancy test (negative human coriogonadotropine (hCG) urine test).
* The subject gives informed consent.

Exclusion Criteria:

* • Pregnant or lactating women.

  * Women of childbearing age (period of time from menarche to postmenopausal status, defined as 12 months absence of menstruation without other medical cause) who do not follow the contraceptive methods recommended by the Clinical Trial Facilitation Group (CTFG) (https://www.hma.eu/fileadm/dateien/Human_Medicines/01): Hormonal contraceptives associated with ovulation inhibitors, intrauterine devices, surgical methods (tubal ligation, vasectomy), abstinence, and barrier methods.
  * Body weight ≤ 60 kg.
  * Presence of liver disease (patients with elevated liver enzyme levels alanine aminotransferase (ALT) / aspartate aminotransferase (AST)> 2x the upper limit of normal, or total bilirubin> 1.5 ULN).
  * Thrombopenia (<100.000 platelets/mL).
  * Be on treatment with other anticoagulants (heparins) or antiplatelet drugs.
  * Be treated with enzyme inhibitors (such as azole antifungals or HIV protease inhibitors) or enzyme inducers (such as rifampin, phenobarbital, carbamazepine, or phenytoin) of CYP3A4 (Cytochrome P450 3A4 oxidase ).
  * History of bleeding episode in the last month.
  * Presence of clinical or analytical alterations not attributable to the stage of kidney disease
  * Participation in another clinical trial of pharmacological treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2021-05-20 (Actual); Primary Completion 2022-12-15 (Actual); Study Completion 2022-12-15 (Actual)

PRIMARY OUTCOMES:
Blood plasma concentrations of Apixaban before, during and after renal replacement therapy | 28 days
  Determine the plasma concentrations of apixaban before, during and after renal replacement therapy (hemodialysis and hemodiafiltration)

SECONDARY OUTCOMES:
Urine plasma concentrations of Apixaban before, during and after renal replacement therapy | 28 days
  Study the elimination of apixaban in urine (in those patients with residual diuresis)
Anti-Factor Xa activity of apixaban (heparin activity (IU/mL)) | 28 days
  Determine the heparin activity (IU/mL) before, during and after renal replacement techniques (hemodialysis and hemodiafiltration)
Number of patients with medical complications with medical complications not directly related to the underlying disease. | 28 days
  To assess the number of patients with medical complications with medical complications not directly related to the underlying disease.
Dyalisate concentrations of Apixaban before, during and after renal replacement therapy | 28 days
  Determine the dyalisate concentrations of apixaban during renal replacement therapy (hemodialysis and hemodiafiltration)
Total number of adverse events. | 28 days
  Total number of adverse events.
Economic impact of anticoagulant treatment with apixaban compared to anticoagulant treatment with coumarins- part 1 | 28 days
  cost of AVK drug
Economic impact of anticoagulant treatment with apixaban compared to anticoagulant treatment with coumarins- part 2 | 28 days
  cost of INR measurements
Economic impact of anticoagulant treatment with apixaban compared to anticoagulant treatment with coumarins- part 3 | 28 days
  incremental cost-effectiveness ratios (ICERs)
Economic impact of anticoagulant treatment with apixaban compared to anticoagulant treatment with coumarins- part 4 | 28 days
  QALY (quality-adjusted life-year)

CONTACTS AND LOCATIONS:
Locations (1):
- Carolina Polo, Barcelona, Spain